CLINICAL TRIAL: NCT01848873
Title: Efficacy of Amlodipine-folic Acid Tablets on Reduction of Blood Pressure and Plasma Homocysteine in Patients With Mild to Moderate Hypertension and Hyperhomocysteinemia ：a Double-blind Randomized Controlled Trial
Brief Title: Efficacy of Amlodipine-folic Acid Tablets on Reduction of Blood Pressure and Plasma Homocysteine
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Ausa Pharmed Co.,Ltd (Industry)
Collaborators: Peking University First Hospital (Other); Chinese PLA General Hospital (Other); Capital Medical University (Other); Fudan University (Other); Ruijin Hospital (Other); Nanchang University (Other); First Affiliated Hospital of Fujian Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); China Medical University, China (Other); Xi'an Jiaotong University (Other); Xuzhou Medical University (Other); Anhui Medical University (Other); Huazhong University of Science and Technology (Other); West China Hospital (Other); Guangdong Provincial People's Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUSA-amlodipine
Record Dates: First submitted 2013-05-04; First posted 2013-05-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Essential Hypertension
Keywords: Hyperhomocysteinemia; Amlodipine-folic acid tablets; Hypertension; MTHFR C677T
MeSH Terms: conditions — Essential Hypertension; Hyperhomocysteinemia; Hypertension | interventions — Amlodipine; Population Groups; Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- amlodipine-FA tablet, low dose group (Experimental): 5mg amlodipine combined with 0.4 mg of folic acid (FA),once daily for 8 weeks.
  Interventions: Drug: amlodipine-FA tablet, low dose group
- amlodipine-FA tablet ,high dose group (Experimental): 5mg amlodipine combined with 0.8 mg of folic acid (FA), once daily for 8 weeks.
  Interventions: Drug: amlodipine-FA tablet ,high dose group
- amolodipine (Active Comparator): 5 mg amlodipine, once daily for 8 weeks.
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — amlodipine 5mg daily
  Other Names: control
  Arms: amolodipine
Drug: amlodipine-FA tablet, low dose group — 5mg amlodipine combined with 0.4 mg of folic acid, daily.
  Other Names: low dose
  Arms: amlodipine-FA tablet, low dose group
Drug: amlodipine-FA tablet ,high dose group — amlodipine 5mg and folic acid 0.8mg daily
  Other Names: high dose
  Arms: amlodipine-FA tablet ,high dose group

SUMMARY:
To evaluate the efficacy of Amlodipine-folic Acid Tablets on reduction of blood pressure and plasma homocystein.

DETAILED DESCRIPTION:
Traditional risk factors are estimated to account for only part of cardiovascular disease (CVD) risk. Non-traditional risk factors such as increased homocysteine concentration are believed to be causally related to CVD. The interactive effect between hypertension and hyperhomocysteinemia on the risk of CVD has received great attention. Methylenetetrahydrofolate reductase (MTHFR) was the main regulatory enzymes for homocysteine metabolism. MTHFR converts 5, 10-methylene-THF into 5-methyl-THF. Polymorphism of MTHFR C677T leads to a reduction in enzyme activity, which may lead to an increased concentration of plasma homocysteine and lower levels of serum folate, particularly in those with low folate intake. In the present study, we sought to assess: (1) the efficacy and safety of Amlodipine-folic Acid Tablets in lowering blood pressure and homocystein in patients with mild to moderate hypertension and hyperhomocysteinemia (hcy≥10μmol/L);(2) if the blood pressure and homocysteine-lowering efficacy of Amlodipine-folic Acid Tablets can be modified by individual methylenetetrahydrofolate reductase (MTHFR) C677T polymorphisms.

In all, about 756 patients with mild or moderate hypertension and hyperhomocysteinemia will be recruited from about 18 hospitals in different Chinese regions. All hospitals are certified as clinical pharmacology centers by the State Food and Drug Administration (SFDA) in China. Eligible subjects are randomly and double-blindly assigned to one of the three treatment groups: 1) amlodipine tablet (5 mg, control group); 2) amlodipine-folic acid tablet (5mg amlodipine combined with 0.4 mg of folic acid, low FA group); or 3) amlodipine-folic acid tablet (5 mg amlodipine combined with 0.8 mg of folic acid, high FA group), once daily for 8 weeks.

The allocation of participants was programmed by an independent statistical coordinating center, encrypted, and sent to each study center. Tablet containers were labeled only with the name of the trial and the allocated concealment number. The participants, care partners, and all staff directly involved in the trial were blinded to interventions during the period of the trial.

Demographic and clinical information were obtained at baseline. Blood pressure was examined at baseline and every two weeks for a total period of 8 weeks. Blood homocysteine and folate concentrations were examined at baseline and at 4 and 8 weeks of the trial. MTHFR C677T genotypes were determined for each study subject.

All analyses will be performed according to the principle of intention to treat.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years;
2. Seated systolic blood pressure (SBP) between 140 mmHg and 180 mmHg and/or seated diastolic blood pressure between 90 mmHg and 110 mmHg;
3. Plasma homocysteine ≥10umol/L；
4. Signed the written informed consent.

Exclusion Criteria:

1. Pregnant women or women within lactation period;
2. Hypersensitive to calcium channel blocker (CCB) or folic acid;
3. Easily hypersensitiveness
4. Diagnosed secondum hypertension or skeptical secondum hypertension;
5. Severe hypertension (sedentary systolic blood pressure≥180mmHg and/or sedentary diastolic blood pressure≥110mmHg)
6. Severe diseases:

   1. Cardiovascular system:
   2. Diagnosed cardia insufficiency (NYHAⅢ level and higher); Hypertrophic obstructive cardiomyopathy (HOCM);Clinical significantly valvular disease of the heart (VDH);Acute coronary syndrome or coronary artery interventional therapy or coronary artery bypass graft within three months; Severe arrhythmia such as atrial flutter, atrial fibrillation, atrioventricular block above Ⅱ level, et al;
   3. Alimentary system:
   4. Active virus hepatitis; Any of alanine aminotransferase (ALT), aspartate aminotransferase (AST), galactosylhydroxylysyl glucosyltransferase (GGT), alkaline phosphatase (ALP), total bilirubin (TBIL), direct bilirubin (DB) was above 2 times of it's normal value upper limit, albumin (ALB) ≤30g/L;Stomach bulk resect and gastrojejunostomy, stomach intestine malabsorption;
   5. Urinary system:
   6. Serum creatinine≥200μmol/L ; Diagnosed stenosis of renal artery, solitary kidney, renal transplantation;
   7. Endocrine system:
   8. Type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus (fasting glucose≥11.1mmol/L); Diagnosed and uncontrolled hyperthyrosis;
   9. Respiratory system:
   10. Pulmonary heart disease , chronic obstructive lung disease;
   11. Nervous or psyche system:
   12. Transient ischemia attach (TIA) or stoke within 3 months; Severe peripheral nerve or vegetative nerve functional disturbance; Psyche or nervous system dysfunction;Drugs or alcohol dependence.
   13. Others:
   14. Malignant tumor, malnutrition, haematogenesis dysfunction, et al;
7. Obvious signs or abnormal laboratory examination;
8. Taking other antihypertensive drugs and unwilling to stop;
9. Taking folic acid or other Vitamin B groups unwilling to stop.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Combined effective rate of blood pressure and plasma homocysteine reduction | Blood pressure was examined at baseline and every 2 weeks for a total period of 8 weeks. Blood homocysteine concentrations were measured at baseline and at 4 and 8 weeks of the trial.

SECONDARY OUTCOMES:
Blood pressure reduction or plasma homocysteine reduction | Blood pressure was examined at baseline and every two weeks for a total period of 8 weeks. Blood homocysteine concentrations was examined at baseline and at 4 and 8 weeks of the trial.

OTHER OUTCOMES:
24-hour ambulatory blood pressure | 24-hour ambulatory blood pressure were examined at baseline and at 8 weeks of the trial in 96 participants.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, MD, Principal Investigator — Peking University First Hospital, Beijing, CHINA
Locations (16):
- China (16):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Anzhen Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - First Affiliated Hospital of Harbin Medical University, Haibin, Heilongjiang
  - Union Hospital, Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of the School of Medicine, Xi'an Jiaotong University, Xi’an, Shanxi
  - West China School of Medicine, West China Hospital ,Sichuan University, Chengdu, Sichuan
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang